CLINICAL TRIAL: NCT06807983
Title: Impact of a Management Strategy for Acute Dyspnea in Elderly Subjects Based on the Use of Lung and Cardiac Ultrasonography
Brief Title: LUng and Cardiac Ultrasound for REspiratory Distress in ElDerly
Acronym: LUCREED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RC31/23/0386; 2024-A01678-39 (Other: ID-RCB)
Record Dates: First submitted 2025-01-22; First posted 2025-02-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Dyspnea; Respiratory Distress Syndrome
Keywords: Elderly; Point-of-Care Ultrasound; Respiratory Distress Syndrom; Dyspnea
MeSH Terms: conditions — Dyspnea; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: stepped-wedge randomized
Who Masked: Outcomes Assessor
Masking Description: Diagnostic classification and therapeutic adequacy or inadequacy will be established by expert appraisal of the files by 2 experts (a cardiologist and a pulmonologist ) blind to the results of the clinical ultrasound and the the other expert.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clinical ultrasound (Experimental): diagnostic strategy based on the protocolized implementation of clinical lung and cardiac ultrasonography, with a proposed diagnostic and therapeutic focus based on the results.
  Interventions: Diagnostic Test: diagnostic strategy based on lung and cardiac ultrasonography
- standard care (No Intervention): diagnostic and therapeutic strategy based on the usual practices of the department and the clinician

INTERVENTIONS:
Diagnostic Test: diagnostic strategy based on lung and cardiac ultrasonography — cardiopulmonary ultrasound performed by the emergency physician, immediately at patient's bed
  Arms: clinical ultrasound

SUMMARY:
Prospective trial to evaluate the impact on the initial therapeutic inadequacy of a management strategy for acute dyspnea in the elderly based on the use of lung and cardiac ultrasonography.

DETAILED DESCRIPTION:
Acute dyspnea is a frequent and serious reason of admission in Emergency Department (ED), with a one-month mortality close to 16%. It is difficult to diagnose in the initial assessment phase since the cause of this symptom can vary (cardiological, pulmonary, infectious, etc.) and the symptoms can be misleading. This difficulty in diagnosing delays the implementation of appropriate therapeutic management even as the timeliness of management is associated with a reduction in mortality. These issues are particularly important in the elderly.

Lung and cardiac ultrasonography performed by the emergency physician, immediately available at the patient's bedside, could reduce the diagnostic and therefore therapeutic delay.

However, the impact of a diagnostic strategy based on lung and cardiac ultrasonography in dyspneic elderly subjects has not been evaluated.

Patients will be randomized in two groups : "standard of care" or "clinical ultrasound" group. Treatments initiated in Emergency Department (ED) will be noted to be compared to final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will be aged over 65 years, affiliated with the French social security system, and presenting to the ED with acute dyspnea (onset <14 days) accompanied by severity signs before or at triage (respiratory rate ≥22 and SpO2 <92% on room air). The enrolling emergency physician (EP) must be the patient's treating physician and must be trained in LuCUS. Written informed consent from the patient or their legal representative is required for inclusion

Exclusion Criteria:

dyspnea secondary to thoracic trauma, dyspnea clearly related to COVID-19, known pulmonary fibrosis or lung cancer, prior administration of specific treatment for dyspnea before inclusion, immediate need for endotracheal intubation, patients identified as being at end-of-life, and individuals under legal guardianship or deprived of liberty.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
therapeutic inadequacy | Hour 1
  therapeutic inadequacy between initiated emergency treatments and the final diagnosis made by expert opinion

SECONDARY OUTCOMES:
correct diagnosis | emergency department discharge (up to hour 4)
  correct diagnosis at the emergency department discharge (compared with final diagnosis made by expert opinion)
duration of emergency department stay | emergency department discharge (up to hour 4)
  duration in emergency department (in hours)
Post-emergency hospital stay | Day 30
  duration in Post-emergency hospital department: in medicine/surgery/obstetrics or follow-up and rehabilitation care (in days)
Number of days alive outside hospital between D0 and D30 | Day 30
  Number of days alive outside hospital between D0 and D30
Care cost | Day 30
  Care cost - Direct and indirect medical cost looking at French social security spendings for patients

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric BALEN, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balen F, Hebrard M, Delmas C, Dubucs X, Noel-Savina E, Costa N, Shourick J; LUC REED investigators; and the LUC REED investigators. Lung and cardiac ultrasound for respiratory distress in the elderly: study protocol of the LUC REED stepped-wedge cluster randomised trial. BMJ Open. 2025 Aug 16;15(8):e104715. doi: 10.1136/bmjopen-2025-104715. PMID 40819865